CLINICAL TRIAL: NCT04334694
Title: Pomeranian atRial flOw reguLatOr iN conGestive hEart failuRe (PROLONGER) Trial
Brief Title: Atrial Flow Regulator in Heart Failure
Acronym: PROLONGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szpitale Pomorskie Sp. z o. o. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01/2020/W
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Congestive Heart Failure
Keywords: atrial flow regulator; heart failure; interatrial shunting
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: All eligible patients will undergo detailed screening using echocardiography, impedance cardiography and right heart catheterization prior to AFR implantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrial flow regulator (Other): In this arm, patients who have elevated left ventricle filling pressures get (Occlutech® AFR device) and optimal therapy for Heart failure (HF).
  Interventions: Device: Atrial flow regulator (Occlutech® AFR device)

INTERVENTIONS:
Device: Atrial flow regulator (Occlutech® AFR device) — Atrial septostomy followed by implantation of AFR.

SUMMARY:
The aim of the study is to assess invasive and non-invasive parameters that may predict clinical improvement in patients with congestive heart failure after implantation of Occlutech® Atrial flow regulator (AFR) device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic heart failure (HF) in NYHA class III or IV ambulatory
* Optimal medical therapy of HF according to European Society of Cardiology (ESC) guidelines for last 6 months
* Hospitalization because of HF decompensation in last 12 months
* Absence of significant valvular disease requiring cardiac surgery
* Life expectancy ≥ 1 year
* Written informed consent obtained from the patient
* Left ventricle ejection fraction (LVEF) ≥ 15%
* Elevated left heart filling pressures:

  1. Pulmonary artery wedge pressure (PAWP) at rest > 15 mmHg or
  2. PAWP > 25 mmHg during hand grip test

Exclusion Criteria:

* Participation in another clinical trial in last 30 days
* Acute infection or sepsis
* Severe coagulation disorder
* Allergy to nickel or titanium
* Severe peripheral artery disease disabling 6 minutes walk test
* Allergy to antiplatelet drugs, oral anticoagulants or heparin
* Contraindication to trans-oesophageal echocardiography (TEE)
* Pregnancy
* Atrial septal defect (ASD) or presence of atrial septal occluder
* Severe patent foramen ovale (PFO) with significant left to right shunt in rest
* Intracardiac thrombus
* Acute coronary syndrome or Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG) in last 6 months
* Severe pulmonary hypertension:

  1. Right atrial pressure ≥ PAWP (measured in right heart catheterization)
  2. Right atrial pressure > 20 mmHg (measured in right heart catheterization)
* Planned heart transplantation
* Transient ischemic attack or stroke within last 6 months
* Cardiac resynchronisation therapy (CRT) within last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 12 months
  Increase in 6 minutes walk test distance

SECONDARY OUTCOMES:
Clinical improvement II | 12 months
  Reduction in New York Heart Association (NYHA) class
Device related adverse event | 12 months
  Device migration, embolization, device related thrombus, shunt occlusion, need for device removal

OTHER OUTCOMES:
Pulmonary artery wedge pressure (PAWP) at rest | 30 days after AFR
  Reduction of PAWP at rest
Pulmonary artery wedge pressure (PAWP) during handgrip test | 30 days after AFR
  Reduction of PAWP during handgrip test
KCCQ-12 | 12 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Clinical adverse event | 12 months
  Cardiac mortality
Clinical adverse event II | 12 months
  Rehospitalization for HF decompensation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Lewicki, MD,PhD, Principal Investigator — Kashubian Cardiovascular Center; University Center for Cardiology
Locations (1):
- Kashubian Cardiovascular Center, Wejherowo, Poland

IPD SHARING:
Plan to Share IPD: Yes
The following data will be available:
  * echocardiography reports
  * right heart catheterization reports
  * clinical and demographic data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after completion of the study.
Access Criteria: The data will be shared on personal request for review process.